CLINICAL TRIAL: NCT00410514
Title: A Phase 2, Randomized, Double-blind, Parallel Group, Placebo Controlled, Multi-center Study to Evaluate the Urodynamics and Safety of YM178 in Male Subjects With Lower Urinary Tract Symptoms (LUTS) and Bladder Outlet Obstruction (BOO)
Brief Title: A Study of Mirabegron (YM178) in Men With Lower Urinary Tract Symptoms (LUTS) and Bladder Outlet Obstruction (BOO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 178-CL-060
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2012-09

CONDITIONS: Lower Urinary Tract Symptoms; Bladder Outlet Obstruction
Keywords: Beta-3 Receptor Agonist; YM178; Men; Lower Urinary Tract Symptoms; Bladder Outlet Obstruction
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder Neck Obstruction; Multiple Endocrine Neoplasia Type 1 | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received matching mirabegron placebo tablets orally once daily for 12 weeks.
  Interventions: Drug: Placebo
- Mirabegron 50 mg (Experimental): Participants received 50 mg mirabegron tablets orally once daily for 12 weeks.
  Interventions: Drug: Mirabegron
- Mirabegron 100 mg (Experimental): Participants received 100 mg mirabegron tablets orally once daily for 12 weeks.
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — oral
  Other Names: YM178; Myrbetriq
  Arms: Mirabegron 100 mg; Mirabegron 50 mg
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
This study examined the safety, tolerability, and efficacy of mirabegron (YM178) compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men 45 years of age or older
* Documented bladder outlet obstruction

Exclusion Criteria:

* History of urinary retention
* Symptomatic and recurrent urinary tract infection (UTI)

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (25):
- United States (15):
  - Tuscon, Arizona
  - Atherton, California
  - Culver City, California
  - Fresno, California
  - San Diego, California
  - Torrance, California
  - Middlebury, Connecticut
  - Tallahassee, Florida
  - Des Moines, Iowa
  - Shreveport, Louisiana
  - Watertown, Massachusetts
  - Garden City, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Virginia Beach, Virginia
- Canada (10):
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Saint John, New Brunswick
  - Halifax, Nova Scotia
  - Kitchener, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Sherbrooke, Quebec

REFERENCES:
- [Background] Nitti VW, Rosenberg S, Mitcheson DH, He W, Fakhoury A, Martin NE. Urodynamics and safety of the beta(3)-adrenoceptor agonist mirabegron in males with lower urinary tract symptoms and bladder outlet obstruction. J Urol. 2013 Oct;190(4):1320-7. doi: 10.1016/j.juro.2013.05.062. Epub 2013 May 30. PMID 23727415

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Started | 65 | 70 | 65
Safety Analysis Set (SAF) | 65 (All patients who received at least 1 dose of double-blind study drug.) | 70 (All patients who received at least 1 dose of double-blind study drug.) | 65 (All patients who received at least 1 dose of double-blind study drug.)
Full Analysis Set (FAS) | 63 (SAF patients with both Qmax & PdetQmax measurements at baseline and 1 or both measured postbaseline.) | 64 (SAF patients with both Qmax & PdetQmax measurements at baseline and 1 or both measured postbaseline.) | 58 (SAF patients with both Qmax & PdetQmax measurements at baseline and 1 or both measured postbaseline.)
Completed | 63 | 67 | 58
Not Completed | 2 | 3 | 7
Not completed — Adverse Event | 2 | 2 | 2
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Non-compliant with study procedures | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg | Total
Number analyzed (Participants) | 65 | 70 | 65 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (8.43) | 64.1 (8.82) | 62.6 (9.92) | 62.7 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 65 | 70 | 65 | 200
Race/Ethnicity, Customized [Number; unit: participants]
  White | 56 | 60 | 59 | 175
  Black or African American | 6 | 6 | 4 | 16
  Asian | 1 | 3 | 2 | 6
  American Indian or Alaskan native | 1 | 0 | 0 | 1
  Other | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment in Maximum Flow Rate (Qmax)
Description: Maximum urinary flow rate (Qmax) was measured by the Investigator using cystometry and was sent to an independent central reading center for review and interpretation.
  Least squares means (LSM) were derived from an analysis of covariance (ANCOVA) model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Week 12
Population: The Full Analysis Set included all patients who received at least 1 dose of double-blind study drug & had both Qmax & PdetQmax measurements at Baseline & 1 or both at any postbaseline on-treatment visit. Data include the last on-treatment assessment for patients who did not complete the Week 12 visit.
Measure: Least Squares Mean (Standard Error); unit: mL/sec
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 58
mL/sec | -0.33 (0.370) | 0.07 (0.366) | 0.30 (0.388)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50 mg; The study was designed to show non-inferiority of mirabegron compared to placebo for both primary outcome measures. The comparison between mirabegron 50 mg and placebo was conducted first. If non-inferiority was demonstrated in this comparison, mirabegron 100 mg was compared to placebo. However, if the first comparison did not demonstrate non-inferiority, no further comparison was made. This procedure maintained the overall type I error of one-sided 2.5%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was -3 mL/sec for Qmax. Mirabegron was considered non-inferior to placebo for Qmax if the lower limit of the 2-sided 95% confidence interval (CI) for the difference from placebo was greater than -3 mL/sec; ANCOVA; LS Mean Difference = 0.40, 95% CI 2-sided [-0.63 to 1.42] — Treatment groups were compared using ANCOVA with pooled center and treatment as factors and the baseline value as a covariate. Centers with less than 12 patients were pooled before the analysis
Statistical Analysis 2: Comparison: Placebo vs Mirabegron 100 mg; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; LS Mean Difference = 0.62, 95% CI 2-sided [-0.43 to 1.68] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline to End of Treatment in Bladder Contractile Index (BCI)
Description: The Bladder Contractile Index (BCI) is a value used to measure the degree of contractility. BCI was calculated using the following formula:
  BCI = pdetQmax + 5Qmax.
  Strong contractility is a BCI > 150, normal contractility is a BCI of 100-150 and weak contractility is a BCI of < 100.
  Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 57
Scores on a scale | 1.25 (3.363) | -2.60 (3.324) | 2.51 (3.567)

3. Primary Outcome: Change From Baseline to End of Treatment in Detrusor Pressure at Maximum Flow Rate (PdetQmax)
Description: Detrusor pressure at maximum urinary flow rate (PdetQmax) was measured by the Investigator using cystometry and was sent to an independent central reading center for review and interpretation.
  Least squares means (LSM) were derived from an analysis of covariance (ANCOVA) model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cmH2O
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 57
cmH2O | 2.92 (2.906) | -3.03 (2.872) | 1.53 (3.086)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50 mg; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 15 cmH2O for PdetQmax. Mirabegron was considered non-inferior to placebo for PdetQmax if the lower limit of the 2-sided 95% confidence interval (CI) for the difference from placebo was less than 15 cmH2O; ANCOVA; LS Mean Difference = -5.94, 95% CI 2-sided [-13.98 to 2.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Mirabegron 100 mg; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; ANCOVA; LS Mean Difference = -1.39, 95% CI 2-sided [-9.73 to 6.96] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline to End of Treatment in Bladder Voiding Efficiency (BVE)
Description: Bladder Voiding Efficiency (BVE) is a product of bladder contractility against the urethral resistance and is measured according to the degree of bladder emptying. BVE is expressed as a percentage and is calculated using the formula:
  Bladder Voiding efficiency = (Voided volume x 100)/maximum cystometric capacity.
  A higher number indicates a higher voiding efficiency. Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent voiding efficiency
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 62 | 64 | 58
Percent voiding efficiency | -3.01 (3.163) | -5.49 (3.093) | 2.06 (3.277)

5. Secondary Outcome: Change From Baseline to Weeks 1, 4, 8, 12 and End of Treatment in Postvoid Residual Volume (PVR)
Description: Healthy micturitions (urinations) result in complete emptying of the bladder. Post Void Residual (PVR) is the volume of urine retained after voiding and was assessed using abdominal ultrasound. An increasing PVR over time is an indicator of abnormal bladder function or detrusor decompensation.
  Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 4, 8 and 12
Population: The Safety Analysis set included all participants who received at least one dose of study drug. End of treatment (EOT) analysis includes the last assessment for patients who did not complete the Week 12 visit; N indicates the number of patients included at each time point.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 65 | 70 | 65
mL
  Change from Baseline at Week 1 [N=63; 66; 63] | -8.10 (6.512) | -2.93 (6.316) | 0.51 (6.480)
  Change from Baseline at Week 4 [N=63; 67; 63] | 1.08 (6.734) | -1.03 (6.506) | 8.63 (6.702)
  Change from Baseline at Week 8 [N=62; 67; 61] | -9.92 (6.922) | 5.11 (6.621) | -3.71 (6.972)
  Change from Baseline at Week 12 [N=59; 63; 57] | 4.65 (11.598) | 21.13 (11.235) | 33.22 (11.822)
  Change from Baseline at EOT [N=64; 70; 65] | 0.55 (10.702) | 17.89 (10.190) | 30.77 (10.598)

6. Secondary Outcome: Safety Assessed by Adverse Events (AEs), Electrocardiogram (ECG), Vital Signs, Physical Exam and Laboratory Tests
Description: Abnormal laboratory parameters, vital signs or ECG data were defined as AEs if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study medication or was clinically significant. A serious AE was an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, was life-threatening, required or prolonged hospitalization or was considered medically important. AEs were assessed by the Investigator for intensity as mild, moderate or severe and for causal relationship to study drug.
Time Frame: From first dose to within 30 days after last dose of double blind study medication (up to 16 weeks).
Population: The Safety Analysis set included all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 65 | 70 | 65
participants
  Adverse events | 28 | 28 | 34
  Mild intensity adverse events | 17 | 16 | 20
  Moderate intensity adverse events | 7 | 10 | 14
  Severe intensity adverse events | 4 | 2 | 0
  Drug-related adverse events | 8 | 5 | 11
  Serious adverse events | 0 | 0 | 0
  AEs leading to study drug discontinuation | 2 | 1 | 2
  Deaths | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline to Weeks 1, 4, 8, 12 and End of Treatment in International Prostate Symptoms Score (IPSS) Total Score
Description: The IPSS is a validated global questionnaire used to assess the degree of "bother" from benign prostatic hyperplasia symptoms and is based on the answers to 7 questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 4, 8 and 12
Population: The Full Analysis Set included all patients who received at least 1 dose of double-blind study drug & had both Qmax & PdetQmax measurements at baseline & 1 or both at any postbaseline on-treatment visit. End of treatment (EOT) includes the last on-treatment assessment for patients who didn't complete Week 12; N is the number of patients included.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 58
scores on a scale
  Change from Baseline at Week 1 [N=63; 63; 57] | -1.7 (0.47) | -2.4 (0.47) | -1.6 (0.50)
  Change from Baseline at Week 4 [N=63; 62; 58] | -4.0 (0.62) | -5.2 (0.62) | -4.4 (0.66)
  Change from Baseline at Week 8 [N=62; 63; 56] | -5.0 (0.68) | -6.3 (0.68) | -5.3 (0.73)
  Change from Baseline at Week 12 [N=58; 61; 52] | -5.2 (0.83) | -6.3 (0.81) | -4.8 (0.89)
  Change from Baseline at EOT [N=63; 64; 58] | -5.0 (0.78) | -6.2 (0.77) | -4.8 (0.83)

8. Secondary Outcome: Change From Baseline to Weeks 1, 4, 8, 12 and End of Treatment in International Prostate Symptoms Score (IPSS) Voiding Score
Description: The IPSS is a validated global questionnaire used to assess the degree of "bother" from benign prostatic hyperplasia symptoms based on the answers to 7 questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The voiding score is the sum of the responses to 4 questions relating to urination (incomplete emptying, intermittency, weak stream and straining) and ranges from 0 to 20 (asymptomatic to very symptomatic).
  Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 58
scores on a scale
  Change from Baseline at Week 1 [N=63; 63; 57] | -0.9 (0.33) | -1.0 (0.33) | -0.5 (0.35)
  Change from Baseline at Week 4 [N=63; 62; 58] | -2.3 (0.41) | -2.5 (0.41) | -2.1 (0.43)
  Change from Baseline at Week 8 [N=62; 63; 56] | -3.0 (0.44) | -3.1 (0.43) | -2.7 (0.47)
  Change from Baseline at Week 12 [N=58; 61; 52] | -3.0 (0.55) | -2.9 (0.53) | -2.3 (0.58)
  Change from Baseline at EOT [N=63; 64; 58] | -2.8 (0.52) | -2.9 (0.51) | -2.4 (0.54)

9. Secondary Outcome: Change From Baseline to Weeks 1, 4, 8, 12 and End of Treatment in International Prostate Symptoms Score (IPSS) Storage Symptom Score
Description: The IPSS is a validated global questionnaire used to assess the degree of "bother" from benign prostatic hyperplasia symptoms based on the answers to 7 questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The storage symptom score is the sum of the responses to 3 questions relating to storage symptoms (frequency, urgency and nocturia) and ranges from 0 to 15 (asymptomatic to very symptomatic).
  Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 58
scores on a scale
  Change from Baseline at Week 1 [N=63; 63; 57] | -0.7 (0.25) | -1.4 (0.25) | -1.0 (0.26)
  Change from Baseline at Week 4 [N=63; 62; 58] | -1.7 (0.31) | -2.6 (0.31) | -2.3 (0.33)
  Change from Baseline at Week 8 [N=62; 63; 57] | -2.1 (0.33) | -3.2 (0.32) | -2.6 (0.35)
  Change from Baseline at Week 12 [N=59; 61; 52] | -2.2 (0.36) | -3.4 (0.35) | -2.5 (0.39)
  Change from Baseline at EOT [N=63; 64; 58] | -2.2 (0.34) | -3.3 (0.34) | -2.5 (0.36)

10. Secondary Outcome: Change From Baseline to Weeks 1, 4, 8, 12 and End of Treatment in Patient Perception of Bladder Condition (PPBC)
Description: The patient perception of bladder condition (PPBC) asks participants to assess their bladder condition using a 6-point validated Likert scale which ranges from 1 (does not cause me any problems at all) to 6 (causes me many severe problems).
  Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 58
scores on a scale
  Change from Baseline at Week 1 [N=63; 63; 57] | -0.2 (0.10) | -0.3 (0.09) | -0.6 (0.10)
  Change from Baseline at Week 4 [N=63; 62; 58] | -0.3 (0.11) | -0.5 (0.11) | -0.6 (0.12)
  Change from Baseline at Week 8 [N=62; 63; 57] | -0.5 (0.12) | -0.7 (0.12) | -0.9 (0.12)
  Change from Baseline at Week 12 [N=60; 61; 53] | -0.6 (0.13) | -0.9 (0.13) | -0.9 (0.14)
  Change from Baseline at EOT [N=63; 64; 58] | -0.6 (0.13) | -0.9 (0.13) | -0.8 (0.13)

11. Secondary Outcome: Change From Baseline to Weeks 1, 4, 8, 12 and End of Treatment in Mean Number of Micturitions Per 24 Hours
Description: A micturition is any voluntary urination, excluding episodes of incontinence only. The mean number of micturitions per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 58
micturitions
  Change from Baseline at Week 1 [N=63; 64; 57] | -0.15 (0.295) | -0.58 (0.291) | -0.48 (0.311)
  Change from Baseline at Week 4 [N=63; 64; 58] | -0.36 (0.333) | -0.90 (0.328) | -1.36 (0.347)
  Change from Baseline at Week 8 [N=62; 63; 57] | -0.61 (0.337) | -1.32 (0.333) | -1.41 (0.352)
  Change from Baseline at Week 12 [N=62; 63; 54] | -0.27 (0.322) | -1.33 (0.318) | -1.23 (0.348)
  Change from Baseline at EOT [N=63; 64; 58] | -0.31 (0.317) | -1.35 (0.313) | -1.37 (0.331)

12. Secondary Outcome: Change From Baseline to Weeks 1, 4, 8, 12 and End of Treatment in Mean Number of Urgency Episodes With Urgency Severity ≥ 3 Per 24 Hours
Description: For each micturition and/or incontinence episode in the 3 days preceding the clinic visit, participants rated the degree of associated urgency (the sudden compelling desire to pass urine, which is difficult to defer) according to the following scale: 0: No Urgency, felt no need to empty my bladder but did so for another reason; 1: Mild Urgency, could postpone passing water for as long as necessary; 2: Moderate Urgency, could postpone passing water for a short while; 3: Severe Urgency, could not postpone passing water; 4: Urge Incontinence, leaked before reaching the toilet.
  Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Urgency episodes
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 58
Urgency episodes
  Change from Baseline at Week 1 [N=63; 64; 57] | 0.09 (0.256) | -0.81 (0.253) | -0.60 (0.271)
  Change from Baseline at Week 4 [N=63; 64; 58] | -0.11 (0.284) | -1.13 (0.281) | -0.95 (0.298)
  Change from Baseline at Week 8 [N=62; 63; 57] | -0.35 (0.288) | -1.43 (0.285) | -0.98 (0.302)
  Change from Baseline at Week 12 [N=62; 63; 54] | -0.33 (0.295) | -1.65 (0.292) | -0.90 (0.320)
  Change from Baseline at EOT [N=63; 64; 58] | -0.33 (0.290) | -1.60 (0.287) | -0.93 (0.304)

13. Secondary Outcome: Change From Baseline to Weeks 1, 4, 8, 12 and End of Treatment in Mean Number of Incontinence Episodes Per 24 Hours
Description: The mean number of incontinence episodes (the involuntary leakage of urine) per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 4, 8 and 12
Population: Full Analysis Set included all patients who received at least 1 dose of double-blind study drug & had both Qmax & PdetQmax measurements at Baseline & 1 or both at any postbaseline on-treatment visit. The analysis only includes patients with >0 incontinence episodes at baseline. End of treatment (EOT) includes patients who didn't complete Week 12.
Measure: Least Squares Mean (Standard Error); unit: Incontinence episodes
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 58
Incontinence episodes
  Change from Baseline at Week 1 [N=9; 18; 13] | -1.16 (0.561) | -0.18 (0.386) | -0.97 (0.516)
  Change from Baseline at Week 4 [N=9; 18; 13 | -0.99 (0.638) | -0.42 (0.439) | -1.60 (0.586)
  Change from Baseline at Week 8 [N=9; 17; 13] | -0.77 (0.558) | -0.70 (0.396) | -2.31 (0.513)
  Change from Baseline at Week 12 [N=9; 17; 13] | -0.98 (0.528) | -0.91 (0.374) | -2.03 (0.485)
  Change from Baseline at EOT [N=9; 18; 13] | -0.96 (0.516) | -0.89 (0.355) | -1.98 (0.474)

14. Secondary Outcome: Change From Baseline to Weeks 1, 4, 8, 12 and End of Treatment in Mean Voided Volume Per Micturition
Description: The mean volume voided per micturition was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 58
mL
  Change from Baseline at Week 1 [N=63; 64; 57] | 2.75 (4.580) | 6.71 (4.508) | 10.38 (4.833)
  Change from Baseline at Week 4 [N=63; 64; 58] | 10.25 (4.779) | 12.55 (4.705) | 18.31 (5.001)
  Change from Baseline at Week 8 [N=62; 63; 57] | 4.53 (4.930) | 14.52 (4.859) | 22.83 (5.163)
  Change from Baseline at Week 12 [N=62; 63; 54] | 4.49 (4.610) | 16.62 (4.549) | 16.20 (5.000)
  Change from Baseline at EOT [N=63; 64; 58] | 5.40 (4.608) | 15.82 (4.537) | 15.80 (4.823)

15. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and End of Treatment in International Consultation on Incontinence Questionnaire - Male Lower Urinary Tract Symptom (ICIQ MLUTS) Total Symptom Score
Description: Male lower urinary tract symptoms were assessed by the ICIQ MaleLUTS questionnaire which consists of 13 questions each on a 0-4 scale (larger scores correspond to worse conditions). The total symptom score ranges from 0 to 52.
  Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 58
scores on a scale
  Change from Baseline at Week 4 [N=60; 60; 58] | -2.8 (0.61) | -4.0 (0.61) | -3.5 (0.63)
  Change from Baseline at Week 8 [N=61; 61; 56] | -3.9 (0.65) | -5.1 (0.65) | -4.9 (0.68)
  Change from Baseline at Week 12 [N=58; 60; 53] | -4.2 (0.76) | -4.9 (0.74) | -5.4 (0.80)
  Change from Baseline at EOT [N=62; 61; 58] | -3.9 (0.73) | -4.8 (0.73) | -5.5 (0.75)

16. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and End of Treatment in International Consultation on Incontinence Questionnaire - Male Lower Urinary Tract Symptom (ICIQ MLUTS) Total Bother Score
Description: The degree to which urinary symptoms bothered participants was assessed by the ICIQ MaleLUTS questionnaire which consists of 13 symptom bother questions each on a 0-10 scale (larger scores correspond to worse outcomes). The total bother score ranges from 0 to 130.
  Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 58
scores on a scale
  Change from Baseline at Week 4 [N=58; 53; 56] | -7.5 (2.71) | -13.6 (2.82) | -10.0 (2.75)
  Change from Baseline at Week 8 [N=57; 57; 53] | -11.6 (2.77) | -21.9 (2.76) | -19.3 (2.86)
  Change from Baseline at Week 12 [N=54; 53; 51] | -15.1 (3.32) | -19.3 (3.35) | -17.4 (3.44)
  Change from Baseline at EOT [N=60; 57; 58] | -14.0 (3.15) | -20.1 (3.21) | -18.6 (3.20)

17. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and End of Treatment in International Consultation on Incontinence Questionnaire - Lower Urinary Tract Symptom Quality of Life (ICIQ-LUTSqol) Symptom Score
Description: Quality of life was assessed by the ICIQ-LUTSqol questionnaire which consists of 19 questions each on a 1-4 scale (larger scores correspond to less quality of life). The total symptom score ranges from 19 - 76.
  Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 58
scores on a scale
  Change from Baseline at Week 4 [N=41; 37; 33] | -3.2 (0.97) | -4.1 (1.03) | -3.1 (1.13)
  Change from Baseline at Week 8 [N=39; 36; 31] | -4.8 (1.03) | -6.4 (1.06) | -5.7 (1.18)
  Change from Baseline at Week 12 [N=40; 30;26] | -4.7 (1.11) | -6.9 (1.29) | -5.7 (1.47)
  Change from Baseline at EOT [N=47; 40; 36] | -4.8 (0.95) | -6.9 (1.03) | -5.0 (1.11)

18. Secondary Outcome: Change From Baseline to Weeks 4, 8, 12 and End of Treatment in International Consultation on Incontinence Questionnaire - Lower Urinary Tract Symptom Quality of Life (ICIQ-LUTSqol) Overall Symptom Interference of Life Score
Description: Participants were asked to rate how much their urinary symptoms interfered overall with their everyday life on a scale from 0 (not at all) to 10 (a great deal).
  Least squares means were derived from an ANCOVA model with the pooled study center and treatment as factors and the baseline value as a covariate.
Time Frame: Baseline and Weeks 4, 8 and 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Number analyzed (Participants) | 63 | 64 | 58
scores on a scale
  Change from Baseline at Week 4 [N=61; 62; 58] | -0.4 (0.26) | -1.2 (0.26) | -1.0 (0.27)
  Change from Baseline at Week 8 [N=60; 63; 57] | -0.9 (0.27) | -1.7 (0.26) | -1.7 (0.28)
  Change from Baseline at Week 12 [N=59; 61; 53] | -1.1 (0.30) | -2.1 (0.29) | -1.9 (0.32)
  Change from Baseline at EOT [N=62; 63; 58] | -1.1 (0.29) | -2.0 (0.28) | -1.9 (0.30)

ADVERSE EVENTS:
Time Frame: From first dose to within 30 days after last dose of double blind study medication (up to 16 weeks).
Arm/Group | Placebo | Mirabegron 50 mg | Mirabegron 100 mg
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/70 | 0/65
Other Adverse Events (participants affected / at risk) | 1/65 | 4/70 | 2/65
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Mirabegron 50 mg (N=70) | Mirabegron 100 mg (N=65)
Nasopharyngitis (Infections and infestations) | 1 | 4 | 2

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.